CLINICAL TRIAL: NCT03967951
Title: CT Radiomic Features of Pancreatic Neuroendocrine Neoplasms
Status: Completed | Type: Observational
Sponsor: Francesco De Cobelli (Other)
Responsible Party: Sponsor-Investigator, Francesco De Cobelli, Professor of Radiology, Head of Clinical and Experimental Radiology, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: panNEN
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: Radiomics; Pancretic neuroendocrine neoplasms (panNEN)
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CT radiomic feature evaluation — Radiomic features will be calculated and extracted from all contrast and non-contrast CT-scans. First order features will be evaluated and high order features will be grouped in parent matrices. Parent matrices of second and third order will be chosen and evaluated.
  In the second part, based on the results of inter-correlation of the operator analysis, the most significant radiomic features will be chosen. Morphological and histopathological features will be evaluated will be.
  Histopathology will be performed on a biopsy specimen; percentage of Ki67 and grading will be evaluated.

SUMMARY:
The aim of this study is to quantify inter-observer variability in delineating pancreatic neuroendocrine neoplasm (PanNEN) on Computerized Tomography (CT) images and its impact on radiomic features (RF), subsequently to this determination, to use CT texture analysis to predict, histological characteristics of PanNEN on CT scans.

DETAILED DESCRIPTION:
CT imaging is the most widely used modality for studying radiomic features due to its ability to assess tissue density, shape, texture and size before, during and after therapy. To the best of the investigator's knowledge, the impact of inter-observer delineation variability on the reliability of CT RF for PanNEN patients, including Hounsfield unit (HU) values-, shape-, and texture-based features, has not yet been assessed. One this has been determined, an additional evaluation will be conducted to correlate the morphologically observed images with their histopathological characteristics.

The ultimate potential objective of this research is to identify and predict characteristics of aggressiveness of PanNEN in CT scans.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* pancreatic neuroendocrine neoplasm with intervention and biopsy
* availability of pre-operatory CT scan with or without IV contrast agent- inInstitution from 2009-2017

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Monocentric, retrospective, observational study. Subjects who fulfill the inclusion criteria will be randomly chosen from our Institutional data-base. Thirty patients will be used to evaluate inter-observer variability and forty patients will be used to evaluate histological characteristics on CT-scans with and without contrast agent).
  Imaged based and clinical variables will be used to construct an overall status of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Interobserver variability in delineating panNENs on CT | 6 months
  Asses inter-observer variability on CT- scans (with contrast alone)

SECONDARY OUTCOMES:
Use CT texture analysis to predict, histological characteristics of PanNEN on CT scans | 6 months
  Evaluate histological characteristics on CT-scans with and without contrast agent in a group of subjects

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Deaprtment of Radiology, IRCCS Ospadale San Raffaele, Milan
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belli ML, Mori M, Broggi S, Cattaneo GM, Bettinardi V, Dell'Oca I, Fallanca F, Passoni P, Vanoli EG, Calandrino R, Di Muzio N, Picchio M, Fiorino C. Quantifying the robustness of [18F]FDG-PET/CT radiomic features with respect to tumor delineation in head and neck and pancreatic cancer patients. Phys Med. 2018 May;49:105-111. doi: 10.1016/j.ejmp.2018.05.013. Epub 2018 May 23. PMID 29866335
- [Derived] Benedetti G, Mori M, Panzeri MM, Barbera M, Palumbo D, Sini C, Muffatti F, Andreasi V, Steidler S, Doglioni C, Partelli S, Manzoni M, Falconi M, Fiorino C, De Cobelli F. CT-derived radiomic features to discriminate histologic characteristics of pancreatic neuroendocrine tumors. Radiol Med. 2021 Jun;126(6):745-760. doi: 10.1007/s11547-021-01333-z. Epub 2021 Feb 1. PMID 33523367